CLINICAL TRIAL: NCT06560411
Title: Evaluation of Automatic Expiratory Positive Airway Pressure (Auto-EPAP) for Management of Upper Airway Obstruction During Non-Invasive Ventilation With Vivo 45 LS
Brief Title: Evaluation of Auto-EPAP for Management of Upper Airway Obstruction During Non-Invasive Ventilation
Acronym: Vivo NOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breas Medical, Inc. (Industry)
Collaborators: Veranex, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BMCI-002
Record Dates: First submitted 2024-08-08; First posted 2024-08-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Obesity Hypoventilation Syndrome (OHS); Chronic Obstructive Pulmonary Disease (COPD); Neuromuscular Diseases (NMD)
Keywords: Sleep Apnea; Non-Invasive Ventilation (NIV); Respiratory Failure; Polysomnography; Apnea-Hypopnea Index (AHI); Expiratory Positive Airway Pressure (EPAP)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome; Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Sleep Apnea Syndromes; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The study is a prospective, multicenter, single-blind, randomized, cross-over study design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study subjects will be blinded to the sequence arm that they are randomized to. Investigators and site study staff will be unblinded. The scorer(s) of the polysomnography will be blinded to which therapy is being used for objective determination of the primary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Auto Night One, Manual Night Two (Active Comparator): Will undergo Automatic Expiratory Positive Airway Pressure (EPAP) during Non-Invasive Ventilation in polysomnography (PSG) Night 1; Will undergo Manual EPAP during Non-Invasive Ventilation in PSG Night 2
  Interventions: Device: Non-Invasive Ventilation
- Manual Night One, Auto Night Two (Active Comparator): Will undergo Manual Expiratory Positive Airway Pressure (EPAP) during Non-Invasive Ventilation in polysomnography (PSG) Night 1; Will undergo Auto-EPAP during Non-Invasive Ventilation in PSG Night 2
  Interventions: Device: Non-Invasive Ventilation

INTERVENTIONS:
Device: Non-Invasive Ventilation — Provide continuous or intermittent ventilatory support for the care of individuals who require mechanical ventilation

SUMMARY:
To evaluate the safety and effectiveness of the Automatic Expiratory Positive Airway Pressure (Auto-EPAP) feature versus manual expiratory positive airway pressure (EPAP) in the Vivo 45 LS Ventilator.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to provide written informed consent.
2. Subject is ≥ 18 years old.
3. Subject has documented respiratory failure (e.g. sleep hypoventilation with historical transcutaneous carbon dioxide (PtCO2) increase ≥ 10mmHg) and/or daytime hypercapnia (>45 mmHg).
4. Subject is currently using non-invasive positive pressure ventilation (NIV) for 1 month.
5. Subject has a previously documented apnea-hypopnea index (AHI) ≥ 5/hr.
6. Subject's expiratory positive airway pressure (EPAP) settings were recently (≤ 12 months) reviewed.

Exclusion Criteria:

1. Subject is not compliant on NIV (e.g., < 4 hr./night).
2. Subject is pregnant.
3. Subject is on oxygen therapy ≥ 5 L/min.
4. Subject has an invasive interface (e.g. tracheostomy).
5. Subject has had an acute exacerbation within the last 3 months that resulted in a hospitalization.
6. Subject is acutely ill, medically complicated, or who are medically unstable.
7. Subject in whom NIV therapy is otherwise medically contraindicated.
8. Subject has had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
9. Subjects with untreated, non-obstructive sleep apnea (OSA) sleep disorders, including but not limited to: insomnia, periodic limb movement syndrome, or restless leg syndrome.
10. Subjects who have the following pre-existing conditions: severe bullous lung disease, recurrent pneumothorax or pneumomediastinum, cerebrospinal fluid leak, or recent cranial surgery or trauma.
11. Subject does not comprehend English.
12. Subject is unable or unwilling to provide written informed consent.
13. Subject is physically and/or mentally unable to comply with the protocol.
14. Subject is not suitable to participate in the trial for any other reason in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Exploratory effectiveness endpoint is to evaluate the subject's mean Oxygen Desaturation Index (ODI4%) during each overnight polysomnography assessment. | Up to Five Weeks
  The log of the subject's mean Oxygen Desaturation Index (ODI4%) measured during each overnight polysomnography assessment (i.e., log10 (mean+1)).
Exploratory effectiveness endpoint is to evaluate the log of the subject's mean Apnea Hypopnea Index (AHI) during each overnight polysomnography assessment. | Up to Five Weeks
  The log of the subject's mean Apnea Hypopnea Index (AHI) measured during each overnight polysomnography assessment (i.e., log10 (mean+1)).
The primary safety endpoint is the occurrence of device-related serious adverse events (SADEs). | Up to Five Weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Insomnia and Sleep Institute of Arizona, LLC, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - Delta Waves, Colorado Springs, Colorado
  - Bogan Sleep Consultants, Columbia, South Carolina